CLINICAL TRIAL: NCT06854042
Title: A First-In-Human, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Oral E1018 in Healthy Adult Subjects
Brief Title: A Study of Oral E1018 in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E1018-G000-001; CDMRPPR210253-A (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Malaria; Healthy Participants
Keywords: E1018
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: E1018 or Placebo (Experimental)
  Interventions: Drug: E1018; Drug: Placebo
- Cohort 2: E1018 or Placebo (Experimental)
  Interventions: Drug: E1018; Drug: Placebo
- Cohort 3: E1018 or Placebo (Experimental)
  Interventions: Drug: E1018; Drug: Placebo
- Cohort 4: E1018 or Placebo (Experimental)
  Interventions: Drug: E1018; Drug: Placebo

INTERVENTIONS:
Drug: E1018 — Specified dose on specified days.
Drug: Placebo — E1018 matching placebo on specified days.

SUMMARY:
The primary purpose of the study is to evaluate the safety and tolerability of single ascending oral doses of E1018 in healthy adult participants and to evaluate the pharmacokinetics (PK) of E1018 in plasma and urine after single oral dose administration.

ELIGIBILITY:
Inclusion criteria:

1. Nonsmoking/vaping, male or female, age greater than or equal to (>=) 18 years to less than or equal (<=) 55 years old at the time of informed consent. To be considered nonsmokers, participant must have discontinued smoking/vaping for at least 4 weeks before dosing.
2. Body Mass Index (BMI) >=18 and less than (<) 30 kilogram per square meter (kg/m^2) at Screening.

Exclusion criteria:

1. Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic gonadotropin [β-hCG] (or human chorionic gonadotropin [hCG]) test with a minimum sensitivity of 25 international units per liter (IU/L) or equivalent units of β-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the dose of study drug.
2. Females of childbearing potential. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (that is, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
3. Males who have not had a successful vasectomy (confirmed azoospermia) if their female partners are of childbearing potential and are not willing to use a highly effective contraceptive method, as described below, throughout the study period and for 28 days after study drug discontinuation. If the female partner is pregnant, then males who do not agree to use latex or synthetic condoms throughout the study period and for 28 days after study drug discontinuation. No sperm donation is allowed during the study period and for 28 days after study drug discontinuation. The duration may be expanded further based on the half-life of the study drug calculated in this study.

   • A highly effective method of contraception includes any of the following:
   * total abstinence (if it is their preferred and usual lifestyle)
   * an intrauterine device or intrauterine hormone-releasing system
   * a contraceptive implant
   * an oral contraceptive (the participant's partner must have been on a stable dose of the same oral contraceptive product for at least 28 days before dosing and must agree to stay on the same dose of oral contraceptive throughout the study and for 28 days after study drug discontinuation). It is permissible that if a highly effective method of contraception is not appropriate or acceptable to the participant's partner, then the participant must agree to use a medically acceptable method of contraception, that is, double-barrier methods of contraception such as latex or synthetic condom plus diaphragm or cervical/vault cap with spermicide. The duration of contraception period may be extended based on the half-life of the study drug calculated in this study.
4. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing.
5. Presence of concurrent febrile illness(es) at Screening or Baseline.
6. Any history of surgery that may affect PK profiles of E1018 (example, hepatectomy, nephrectomy, digestive organ resection) or participants who have a congenital abnormality in metabolism at Screening.
7. Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, ECG finding, or laboratory test results that require medical treatment at Screening or Baseline.
8. Left bundle branch block.
9. History of myocardial infarction, active ischemic heart disease, or clinically significant or uncontrolled arrhythmia.
10. Known history of clinically significant drug allergy at Screening.
11. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening.
12. Known to be human immunodeficiency virus (HIV)-positive at Screening.
13. Active viral hepatitis (A, B or C) as demonstrated by positive serology at Screening.
14. History of drug or alcohol dependency or abuse, or those who have a positive urine drug test or breath alcohol test at Screening or Baseline.
15. Currently enrolled in another clinical study or used any investigational drug or device within 30 days or 5 half-lives (whichever is longer) preceding informed consent.
16. Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week of dosing.
17. A history of noncompliance in any previous study or inability to comply with study conduct, as assessed by the investigator.
18. Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Events | Up to Day 20
Number of Participants With Adverse Events (Serious and Non-serious) | Up to Day 20
Number of Participants With Clinically Significant Laboratory Test Results | Up to Day 20
Number of Participants With Clinically Significant Vital Signs Values | Up to Day 20
Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Results | Up to Day 20
AUC(0-t): Area Under the Concentration-time Curve From Zero Time to Time of Last Quantifiable Concentration for E1018 | Up to Day 20
AUC(0-inf): Area Under the Concentration-time Curve From Zero Time Extrapolated to Infinite Time for E1018 | Up to Day 20
Cmax: Maximum Observed Concentration for E1018 | Up to Day 20
Tmax: Time at Which the Highest Drug Concentration Occurs for E1018 | Up to Day 20
t½: Terminal Elimination Phase Half-life for E1018 | Up to Day 20
CL/F: Apparent Total Clearance Following Oral Administration for E1018 | Up to Day 20
Vz/F: Apparent Volume of Distribution at Terminal Phase for E1018 | Up to Day 20
Ae: Cumulative Amount of E1018 Excreted in the Urine | Up to Day 6
Fe: Percent (%) of Administered E1018 Dose Excreted in Urine | Up to Day 6

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.